CLINICAL TRIAL: NCT06805032
Title: Accuracy and Precision of Train-of-Four Ratios Obtained With Acceleromyography and Electromyography in Restricted-Movement Settings in the Absence of Neuromuscular Blocking Drugs
Status: Enrolling by invitation | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, J. Ross Renew, M.D., Principal Investigator, Mayo Clinic
Other Study IDs: 24-011159
Record Dates: First submitted 2025-01-28; First posted 2025-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Cystoscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Procedure without neuromuscular blockade
  Interventions: Other: Observation of EMG and AMG readings

INTERVENTIONS:
Other: Observation of EMG and AMG readings — Simultaneous readings from electromyograph and acceleromyograph

SUMMARY:
The purpose of this research is to compare the performance of acceleromyograph and electromyograph-based quantitative neuromuscular monitors when the arms are tucked for surgical positioning.

ELIGIBILITY:
Inclusion Criteria:

* Patients willing to participate and provide an informed consent.
* Patients undergoing elective surgical procedures that require general anesthesia without use of NMBA agents administered intraoperatively, and tucked arms.
* Anticipated surgery duration < 120 minutes.

Exclusion Criteria:

* Patients with disorders, such as stroke, carpal tunnel syndrome, broken wrist with nerve damage, Dupuytren contracture, or any similar wrist injury.
* Patients with systemic neuromuscular diseases such as myasthenia gravis.
* Patients having surgery that would involve prepping the arm into the sterile field.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective surgery and requiring general anesthesia without administration of neuromuscular blocking agents.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-03-25 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Accuracy and precision | 120 minutes
  Accuracy and precision of train-of-four ratios measured simultaneously by two quantitative neuromuscular monitors every minute among 40 patients undergoing surgery of at least 30 min duration (roughly 1200 measurements) in which the arms are tucked and in the absence of neuromuscular blocking agents. In the absence of neuromusuclar blocking agents, the expected train-of-four ratio is 1.0. Accuracy of each monitor will be assessed by how close measuremetns are to 1.0 while precision will be assessed by the variability of the measured responses in all patients undergoing procedure.

CONTACTS AND LOCATIONS:
Overall Officials: J. Ross Renew, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No